CLINICAL TRIAL: NCT04397003
Title: Phase II Study of a Personalized Neoantigen Vaccine in Combination With Durvalumab (MEDI4736) in Extensive Stage Small Cell Lung Cancer
Brief Title: Personalized Neoantigen Vaccine in Combination With Durvalumab (MEDI4736) in Extensive Stage Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: AstraZeneca (Industry); Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202104143
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoantigen DNA vaccine+durvalumab (Experimental): * Patients will receive durvalumab (1500mg Q3W) in combination with standard of care carboplatin and etoposide for a total of 4 cycles given every 3 weeks
  * Beginning 4 weeks following Cycle 4 of carboplatin/etoposide/durvalumab, patients on will then receive 6 cycles of durvalumab 1500 mg with the polyepitope neoantigen DNA vaccine, both administered once every 4 weeks
  * Patients may then receive durvalumab every 4 weeks until disease progression or drug toxicity
  * Should a delay in vaccine preparation occur, patients will begin durvalumab and the vaccine will be added with the subsequent cycle.
  Interventions: Biological: Neoantigen DNA vaccine; Drug: Durvalumab; Device: TDS-IM v2.0 Device; Procedure: Peripheral blood draws

INTERVENTIONS:
Biological: Neoantigen DNA vaccine — All study injections will be given intramuscularly using an integrated electroporation device (TDS-IM system, PapiVax Biotech). At each vaccination time point, patients will receive two injections of the neoantigen DNA vaccine, one injection into each deltoid or lateralis.
Drug: Durvalumab — -Supplied by AstraZeneca
  Other Names: Imfinzi
Device: TDS-IM v2.0 Device — -Integrated electroporation administration system
Procedure: Peripheral blood draws — -Pre-treatment, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Vaccine Day 1, Vaccine Day 29, Vaccine Day 85, Vaccine Day 141, on even numbers of cycles for durvalumab for one year following completion of vaccine

SUMMARY:
The investigators hypothesize that a personalized neoantigen vaccine combined with durvalumab will improve the progression free survival of patients with extensive state small cell lung cancer (ES-SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive stage small cell lung cancer (ES-SCLC)
* Considered suitable to receive a platinum-based chemotherapy regimen with durvalumab as 1st line treatment for ES-SCLC.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* At least one lesion must be able to be biopsied at the time of enrollment. The site utilized for biopsy cannot be utilized as a target lesion for efficacy measurement.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Life expectancy of at least 12 weeks.
* Body weight > 30 kg.
* Adequate normal organ and marrow function as defined below:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1.0 K/cumm
  * Platelet count ≥ 75 K/cumm
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x IULN unless liver metastases are present, in which case it must be ≤ 5 x IULN
  * Measured creatinine clearance > 40 mL/min or calculated creatinine clearance > 40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
* Adequate cardiac function defined as QTcF < 470 ms on 12-lead ECG.
* Baseline pulse oximetry must be > 92% on room air.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy):
* Male and female patients of reproductive potential must be willing to employ effective birth control from screening to 90 days after the last dose of durvalumab
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable). This includes consent for tumor/normal exome sequencing and dbGaP-based data sharing.

Exclusion Criteria:

* Prior treatment with a PD-1 or PD-L1 inhibitor (including durvalumab).
* A history of other primary malignancy except for:

  * Malignancy treated with curative intent and with no know active disease ≥ 5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Currently receiving any other investigational agents.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
* Any unresolved toxicity NCI CTCAE grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

  * Patients with grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the PI.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the PI.
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
* Major surgical procedure (as defined by the PI) within 28 days prior to the first dose of study drug. Note: local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* History of leptomeningeal carcinomatosis.
* Any known history of brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab or other agents used in the study.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Uncontrolled intercurrent illness including, but not limited to:

  * uncontrolled ongoing or active infection
  * a history of myocarditis or congestive heart failure (as defined by New York Heart Association Functional Classification III or IV)
  * myocardial infarction 6 months prior to study entry
  * uncontrolled hypertension
  * unstable angina pectoris
  * serious uncontrolled cardiac arrhythmia
  * interstitial lung disease (ILD) or a history of ILD/pneumonitis requiring treatment with systemic steriods
  * serious chronic gastrointestinal conditions associated with diarrhea
  * psychiatric illness or social situations that would limit compliance with study requirements, substantially increase the risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug. Note: patients, if enrolled, should not receive live vaccine whilst receiving study drug and up to 30 days after the last dose of study drug.
* History of syncopal or vasovagal episode as determined by medical record and history in the 12 month period prior to enrollment
* Less than 2 acceptable potential injection sites for IM injection and electroporation considering the left and right medial deltoid, and anterolateral quadriceps muscles. A site for injection and electroporation is not acceptable if there is inadequate muscle mass to support at least a 19 mm /0.75 inch injection depth or a skin pinch thickness measurement of >50 mm as assessed using the provided caliper). Eligible injection sites must also have intact lymphoid drainage and be free from tattoos, hypertrophic skin patches, keloids or other skin conditions which could interfere with the administration procedure or subsequent assessment of local reactogenicity. Note: In order to ensure adequate muscle mass for administrations for participants with a weight <65 kg, potentially eligible administration sites are confined to the outer aspect of the upper thigh (left or right vastus lateralis muscle). The left and right medial deltoid are not eligible administration sites for those participants.
* Is an individual in whom the ability to observe possible local site reactions at >2 eligible injection sites (left and right medial deltoid or left and right vastus lateralis muscles) is, in the opinion of the investigator, unacceptably obscured due to a physical condition.
* Has a metal implant or implantable device within the area of the electroporation injection site at >2 of the eligible injection sites.
* Contraindication to intramuscular injections and/or blood draws.
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child.
* Current use of any non-removable electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]. The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* History of primary active immunodeficiency.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

Reconfirmation of Eligibility Prior to Administration of Neoantigen DNA Vaccine:

Inclusion Criteria:

* Eligible to receive durvalumab
* ECOG performance status ≤ 1
* Body weight > 30 kg
* Baseline pulse oximetry must be > 92% on room air

Exclusion Criteria:

* Currently receiving any other investigational agents
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Less than 2 acceptable potential injection sites for IM injection and electroporation considering the left and right medial deltoid, and anterolateral quadriceps muscles. A site for injection and electroporation is not acceptable if there is inadequate muscle mass to support at least a 19 mm /0.75 inch injection depth or a skin pinch thickness measurement of >50 mm as assessed using the provided caliper. Eligible injection sites must also have intact lymphoid drainage and be free from tattoos, hypertrophic skin patches, keloids or other skin conditions which could interfere with the administration procedure or subsequent assessment of local reactogenicity. Note: In order to ensure adequate muscle mass for administrations for participants with a weight <65 kg, potentially eligible administration sites are confined to the outer aspect of the upper thigh (left or right vastus lateralis muscle). The left and right medial deltoid are not eligible administration sites for those participants.
* Individuals in whom the ability to observe possible local site reactions at >2 eligible injection sites (left and right medial deltoid or left and right vastus lateralis muscles) is, in the opinion of the investigator, unacceptably obscured due to a physical condition
* Has a metal implant or implantable device within the area of the electroporation injection site at >2 of the eligible injection sites
* Contraindication to intramuscular injections and/or blood draws
* Current use of any non-removable electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the combination of durvalumab and a neoantigen vaccine as measured by number of participants experiencing adverse events | Through 90 days after completion of treatment (estimated to be 2 years and 3 months)
  -Safety and tolerability will be measured by National Cancer Institute Common Terminology Criteria (NCI CTCAE) v 5.0
Feasibility of combining durvalumab with a neoantigen vaccine as measured by the number of participants that had a vaccine produced for them | Within 24 weeks of the start of consolidation durvalumab
  -Feasibility is defined as the ability to produce a vaccine for 80% of patients enrolled within 24 weeks of the start of consolidation durvalumab.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 12 months
  * PFS is defined as the duration of time from start of durvalumab to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Response conversion rate | Through completion of treatment (estimated to be 2 years)
  -The response conversion rate is defined as the proportion of patients who improve in RECIST v1.1 category subsequent to vaccination.
Duration of response (DOR) | Through completion of treatment (estimated to be 2 years)
  -The duration of response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Overall survival (OS) | Through completion of follow-up (estimated to be 4 years and 3 months)
  -Defined as time from start of durvalumab to death due to any causes

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Ward, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All study data will be shared with the study sponsor and will be available from presentations and upon publication.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu